CLINICAL TRIAL: NCT04425174
Title: The Analgesic Effect of Bilateral Quadratus Lumborum Block and Its Postoperative Implication on Kidney Function in Colorectal Surgery: a Comparative Randomized Control Trial Study With Epidural Anesthesia.
Brief Title: The Analgesic Effect of Quadratus Lumborum Block and Its Postoperative Implication on Kidney Function
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Reham Mustafa Hashim, Clinical Professor, Ain Shams University
Other Study IDs: FMASU R 14/2020
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2021-11-11 (Actual); Status verified 2021-11

CONDITIONS: Anesthesia
Keywords: Quadratus Lumborum block; Renal resistive index; Renal doppler; Epidural anesthesia
MeSH Terms: interventions — Anesthesia, Epidural

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- QL: QL = 30 patients representing the case group receiving QL block.
  Interventions: Procedure: Quadratous lumborum block
- EP: EP = 30 patients representing the control group receiving epidural anesthesia.
  Interventions: Procedure: Epidural anesthesia

INTERVENTIONS:
Procedure: Quadratous lumborum block — Quadratus Lumborum (QL) block is a new technique for analgesia of the abdominal wall muscles. Its mechanism depends on the injection of the local anesthetic agent between the abdominal wall muscles into the thoracolumbar fascia surrounding the Quadratus Lumborum muscle by ultrasound (US) guided technique.
  Groups: QL
Procedure: Epidural anesthesia — Epidural analgesia is a gold standard analgesic technique for the majority of abdominal surgeries, yet it has some limitations in some surgeries as colorectal surgeries due to delayed ambulation due to muscular weakness and postural hypotension.
  Groups: EP

SUMMARY:
Regional anesthesia is frequently used in major surgery in association with general anesthesia to ensure adequate postoperative patient analgesia and to decrease the intra- and postoperative use of systemic analgesic drugs. Epidural analgesia (EP) is considered the standard regional analgesic technique that is widely used in abdominal surgery. Nonetheless, it has some limitations such as in colorectal surgery where complications in the form of muscular weakness, hemodynamic instability, and postural hypotension result in delayed patient ambulation.

For these limitations, peripheral nerve blocks can be considered safer with less incidence of complications compared to the central neuraxial blocks especially with the use of ultrasound (US) as a guide in their techniques. Also, avoidance of the hemodynamic instability that may affect the postoperative kidney function can be considered an important issue in patients with risk for postoperative acute kidney injury (AKI).

One of the latest techniques in the field of regional anesthesia is the quadratus lumborum (QL) block, which is based on US-guided injection of a local anesthetic agent into the thoracolumbar fascia surrounding the QL muscle. Several different approaches were described depending on the injection sites, for example, lateral, posterior, and anterior approaches . According to the ASRA-ESRA Delphi consensus, there was no consensus on naming quadratus lumborum block types where posterior QL had the strongest consensus in abdominal wall analgesia with 71%.

After the QL block, there is evidence that the injectate spreads to the paravertebral space where it blocks the thoracolumbar nerves and the thoracic sympathetic trunk. Because it produces an extensive sensory block leading to adequate postoperative analgesia besides decreasing the systemic analgesic consumption, QL block is now considered an effective regional block that can be used in major abdominal surgery.

40% of the cases diagnosed as having AKI occurred as a postoperative complication. Cardiac surgery carries the highest risk for AKI (18.7%), whereas general surgery comes second (13.2%). The risk factors of developing AKI may be general or causes related to the type and the setting of the surgery.

Fluid depletion is one of the major factors that can occur perioperatively and leads to renal hypoperfusion, with subsequent renal arteriolar changes, attempting to maintain a normal glomerular filtration rate. The sympathetic effects of the neuroendocrine hormones may lead to renal vasoconstriction, aiming to redistribute the blood to the medulla; however, it may lead to renal ischemia.

The renal blood flow can be assessed by a rapid bed-side noninvasive technique, using the renal Doppler resistive index (RI), which is one of the most fundamental parameters assessing renal perfusion, because it reflects the degree of the vascular resistance inside the kidney vascular bed and can be used to assess the modifications and the changes that occur in the renal blood flow.

No previous studies so far discussed the effect of QL block on postoperative creatinine and blood ureal nitrogen (BUN) levels. While, regarding epidural analgesia, multiple articles are investigating the effect of epidural on postoperative kidney function using various indices, such as serum creatinine, BUN, sodium clearance, and urine output. As far as the authors know, this is the first study using the RI renal flow as a comparative parameter between the QL block and EP analgesia.

This study aimed to assess the analgesic efficacy of QL block compared with epidural anesthesia as a primary outcome using the 10-point visual analog scale (VAS), time to first morphine requirement, and 24-hour morphine consumption. Also, to study the effect of both on postoperative kidney function as a secondary outcome using serum creatinine and BUN and renal flow assessment using renal Doppler.

DETAILED DESCRIPTION:
* Study place: Ain Shams University Hospitals.
* Written informed consent will be taken from all patients.
* Patients with an American Society of Anesthesiologists (ASA) physical status I-III, aged between 35 and 65 years were included in this study and scheduled for short colorectal surgery (2-4 hours), such as segmental colectomies and polypectomy using either the sub umbilical incision or laparoscopic technique. Patients with major cardiac or cerebral vascular diseases, bleeding disorders (known contraindication for EP anesthesia and in QL which is considered a deep block), abnormal kidney functions (elevated creatinine, BUN level, or history of renal disease), and neurological disorders were excluded. Patients with known allergy to local anesthetics, puncture site infection, and body mass index (BMI) of >35 kg/m2 were also excluded. Also, patients with intra-operative complications such as hemodynamic instability and unexpected prolonged surgical duration were excluded. Patients who refused to consent to the study were not enrolled, without any discontinuation of their management.

The selected patients were randomized using an automated computer-assisted method (www.randomizer.org), which divided them into 2 groups: the control group (EP) received epidural anesthesia, whereas the study group (QL) received a QL block. The interventions were done by well-experienced anesthesiologists.

Renal Doppler. An experienced radiologist performed the renal Doppler with at least 5 years experience in the doppler field being blinded to the patients' data. A renal Doppler study was performed for both groups preoperatively and postoperatively. Patients were asked to lie supine or in lateral positions. The ultrasound (US) probe was applied to the anterior or midaxillary line with the probe in a transverse direction until the kidney was adequately visualized. The intrarenal and main renal arteries were assessed using color and pulse wave Doppler. The intrarenal arteries assessment was repeated at the upper, mid, and lower pole levels of each kidney. Also, the renal RI of the main renal artery was measured bilaterally. All measurements for each patient were collected and the average RI was calculated. The normal RI is considered when the value was <0.7. The renal Doppler was assessed within 24 hours pre-operative and within 2-3 hours after surgery completion.

Patient preparation. Patients who fasted for 8 hours, with full clinical and laboratory results, were examined for any exclusion criteria with specific concerns with regard to kidney function. 12 hours before the scheduled time for surgery, renal Doppler was performed to measure the renal RI of all patients, before starting to fast for surgery and after adequate hydration was checked, based on his ward fluid chart.

Inside the operating room. The standard monitoring, including electrocardiogram (ECG), oxygen saturation, non-invasive blood pressure, and capnogram for end-tidal carbon dioxide (ETCO2), were applied. Infusion of Ringer's lactate solution (8 mL/kg) was started through a wide bore cannula. IV midazolam 0.05 mg/kg was given as a premedication before the induction of anesthesia by 2 μg/kg fentanyl, 2 mg/kg propofol, and 0.5 mg/kg atracurium. An endotracheal tube was inserted to initiate mechanical ventilation while keeping the ETCO2 in the range of 35-45 mmHg. Anesthesia maintenance was performed with 1.5% isoflurane and oxygen and topped up with IV atracurium 0.5 mg/kg every 20 minutes. The urinary output was followed up using a urinary catheter. IV fentanyl dose of 1 μg/kg was administered, in response to an increase in blood pressure or heart rate of >20% of the baseline measurement. Continuous ECG, blood pressure, and pulse saturation were monitored. To ensure an adequate fluid balance, fluid input, fluid output (urine and third space loss), blood loss, and central venous pressure were recorded. The inhalational anesthetic isoflurane was discontinued at the end of the surgery, followed by the administration of IV neostigmine of 0.05 mg/kg and atropine of 0.02 mg/kg, to reverse the residual neuromuscular block. The trachea was extubated after spontaneous breathing returned.

Epidural analgesia. Epidural analgesia was performed before the induction of general anesthesia by a well-experienced anesthesiologist with at least 5 years experience in local and regional anesthesia. Patients were in a sitting position leaning forward with the legs supported on a chair. Complete skin asepsis with povidone-iodine (7.5%), was applied followed by draping. An 18-gauge Tuohy epidural needle was inserted into the intervertebral space T9-T10, using a vacuum catheter aspiration technique followed by the epidural catheter insertion. The epidural was activated at the end of the operation using 10 mL of 0.25% bupivacaine as a bolus followed by a continuous epidural infusion using 0.125% bupivacaine, at a rate of 6 mL/hour, to be continued for up to 24 hours postoperatively.

QL block technique. A bilateral posterior approach, a US-guided QL block was applied after anesthesia induction by a well-experienced anesthesiologist with at least 5 years experience in local and regional anesthesia, using Honda electronics HS-2100 portable US machine (Honda Electronics CO., LTD, Japan). The patient was in a supine position with a pillow under his back. Povidone-iodine (7.5%) was used to sterilize the area above the iliac crest at the level of the anterior axillary line, followed by draping before the application of a high-frequency superficial probe (9-11 MHz). The probe was adjusted until visualization of the external oblique muscle, the internal oblique muscle, and the transversus abdominis muscle. Then the probe was moved posteriorly until the thoracolumbar fascia covering the QL muscle was visualized. The needle was inserted just above the upper edge of the probe and pierced the muscles until it reached the posterior aspect of the QL muscle. Aspiration was done to ensure that there is no blood and to ensure extravascular injection to avoid the undesirable systemic effect. The correct site was confirmed through saline injection (hydro dissection); 25 mL of 0.25% bupivacaine were injected on each side.

Fluid balance was maintained throughout the operation, using a fluid chart to avoid any hemodynamic instability that might affect the objective of this study.

Postoperative study parameters. Patients were transferred to the intermediate care unit, for continuous observation for 24 hours. A 10-point visual analog scale (VAS) was used to assess pain; with 0 being no pain and number 10 being the worst pain. The VAS score was assessed immediately after patients' transfer from the theater room (0 hours) then 2, 6, 8, 12, 18, and 24 hours postoperative. The following parameters were assessed by a blinded anesthesiologist to the aim of the study:

* The time required for the first morphine dose and the cumulative morphine consumption for 24 hours were recorded as a primary outcome. Morphine was given at a dose of 0.05 mg/kg when the VAS score was >4.
* Postoperative kidney function was assessed using laboratory and US Doppler indices to compare it with the preoperative values, as a secondary outcome. Laboratory tests included serum creatinine and blood urea nitrogen (BUN) and were compared with preoperative values.

ELIGIBILITY:
Inclusion Criteria:

* Patients with an American Society of Anesthesiologists (ASA) physical status I-III.
* Patients aged between 35 and 65 years scheduled for colorectal surgeries.

Exclusion Criteria:

* We will exclude patients with serious cardio-cerebral vascular diseases, neurological disorders, bleeding disorders as QL block is a deep block, allergies to local anesthetics (LAs), infection at the puncture site, body mass index (BMI)> 35kg/m2, history of mental illness, and patients who will not consent to the procedure.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cases will undergo colorectal surgeries
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-08-15 (Actual); Study Completion 2020-09-22 (Actual)

PRIMARY OUTCOMES:
Pain score | 24 hours
  Visual analog score will be assessed post operatively. The score is from 0 to 10 with 0 equal no pain while 10 represents the worst pain.
First morphine dose | 24 hours
  Time of the first morphine dose needed to control post operative pain.
Cumulative morphine dose | 24 hours
  The total amount of morphine used to control post operative pain

SECONDARY OUTCOMES:
Renal doppler | 12 hours
  Measurement of the renal artery resistive index compared to the pre-operative measurements.
Laboratory kidney function | 12 hours
  Assessment of the serum creatinine and blood urea nitrogen (BUN) to be compared with the pre-operative values

CONTACTS AND LOCATIONS:
Overall Officials: Reham M Hashim, Principal Investigator — Faculty of medicine - Ain shams university
Locations (1):
- Reham M. Hashim, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol